CLINICAL TRIAL: NCT05349604
Title: Effect of Garlic Extracts on Changes in Blood Flow Velocity in the Carotid Artery: Randomized, Double-blind, Placebo-controlled Study
Brief Title: Effect of Garlic Extracts on Changes in Blood Flow Velocity in the Carotid Artery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Yong-il Shin, Professor, Pusan National University Yangsan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 04-2020-038
Record Dates: First submitted 2021-06-09; First posted 2022-04-27 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Garlic extracts (Experimental): Take 450mg of Garlic extracts(Food Item Making Report Product Name: Vegetable Extract Powder No. 1905, Item Report No.: 202004980275)
  Interventions: Dietary Supplement: Garlic extracts
- placebo (Placebo Comparator): As a food ingredient that does not affect blood pressure and is harmless to the human body, it is made almost identical in weight and appearance to garlic extract.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Garlic extracts — One intake in total
  Arms: Garlic extracts
Dietary Supplement: Placebo — One intake in total
  Arms: placebo

SUMMARY:
The purpose of this study is to assess the safety and efficacy of Garlic extracts for improving of blood flow velocity in the carotid artery.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults 19 years of age or older as of the screening date
2. Those with no history of treatment for hypertension within the last 3 months
3. A person who voluntarily decides to participate and agrees in writing to abide by the precautions after hearing and fully understanding the detailed explanation of this study

Exclusion Criteria:

1. Those with systolic blood pressure of 160 mmHg or higher or diastolic blood pressure of 100 mmHg or higher
2. Those who have had a stroke, myocardial infarction, percutaneous coronary angioplasty or surgery for coronary angioplasty within the past 6 months
3. Persons with acute and severe cardiovascular diseases such as heart failure, myocardial infarction, and stroke
4. Those with acute/chronic inflammation such as cancer, rheumatic disease, autoimmune disease, gastrointestinal disease, etc.
5. Those who have a history of gastrointestinal diseases (eg Crohn's disease) or gastrointestinal surgery (except simple appendicectomy or hernia surgery) that may affect the absorption of the product for human application testing
6. Persons who have taken prohibited concomitant drugs within the last 3 months
7. Persons with a history of clinically significant hypersensitivity reactions to drugs and health functional foods
8. Those who have received antipsychotic drug treatment within 2 months before the screening test
9. Persons with a history of drug or alcohol abuse
10. Pregnant or lactating women
11. When women of childbearing potential of childbearing potential do not accept the implementation of appropriate contraceptive methods (except for women who have undergone sterilization)
12. Subjects who have participated in health functional food related research or clinical trials within the last 3 months
13. In case the principal investigator judges that it is not appropriate to participate in this study

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-10-27 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Change of peak systolic blood flow velocity in the common carotid arteries | Change of peak systolic blood flow velocity before and after 60 minutes garlic extract intake basis in the experimental group
  Doppler ultrasonography is used for measurement.
Change of end-diastolic blood flow velocity in the common carotid arteries | Change of end-diastolic blood flow velocity before and after 60 minutes garlic extract intake basis in the experimental group
  Doppler ultrasonography is used for measurement.
Change of diastolic and systolic blood pressure | Change of diastolic and systolic blood pressure before and after 60 minutes garlic extract intake basis in the experimental group
  The blood pressure device is measured by IntelliVue MP50® from Philips. When measuring blood pressure, the study subjects should sit comfortably for at least 5 minutes and then take the measurements. The unit is mmHg and is expressed as an integer.
Change of peak systolic blood flow velocity in the internal carotid arteries | Change of peak systolic blood flow velocity before and after 60 minutes garlic extract intake basis in the experimental group
  Doppler ultrasonography is used for measurement.
Change of end-diastolic blood flow velocity in the internal carotid arteries | Change of end-diastolic blood flow velocity before and after 60 minutes garlic extract intake basis in the experimental group
  Doppler ultrasonography is used for measurement.

CONTACTS AND LOCATIONS:
Locations (1):
- Pusan national university Yangsan Hospital, Gyeongsang, Yangsan, South Korea

IPD SHARING:
Plan to Share IPD: No